CLINICAL TRIAL: NCT04140188
Title: Sentinel Lymph Node Biopsy After Nipple Sparing Mastectomy: Prospective Study
Brief Title: SLNB After Nipple Sparing Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Halil KARA, Principal Investigator, Acibadem University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RISA-19-01
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Sentinel Lymph Node Biopsy; Mastectomy, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axilla no touch (Active Comparator): Volunteer patients who did not underwent to SLNB or axillary lymph node dissection during previous NSM
  Interventions: Diagnostic Test: Senti-Scint (99mTc- pertechnetate combined with human albumin)
- Axilla with previous SLNB (Active Comparator): Volunteer patients who has underwent to SLNB but not axillary lymph node dissection during previous NSM
  Interventions: Diagnostic Test: Senti-Scint (99mTc- pertechnetate combined with human albumin)

INTERVENTIONS:
Diagnostic Test: Senti-Scint (99mTc- pertechnetate combined with human albumin) — Senti-Scint will be injected via intradermal route to the breast with history of previous NSM.

SUMMARY:
Sentinel Lymph Node Biopsy (SLNB) after nipple sparing mastectomy (NSM) is controversial. This study aims to investigate feasibility of SLNB with radioisotope method.

DETAILED DESCRIPTION:
Volunteer patients who has underwent to NSM at least more than 6 months prior will be included to the study. Radioisotope will be injected via intradermal route to the breast underwent to NSM patients and lymphoscintigraphy images will be obtained to detect activity in axilla. If hot nodule is detected then it will be concluded that SLNB can be performed after NSM.

ELIGIBILITY:
Inclusion Criteria: NSM with/without SLNB at least 6 months prior to this study -

Exclusion Criteria: previous axillary dissection and active breast cancer

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is rarely seen in male patients and NSM is not performed thus study group consist of female volunteers.
Enrollment: 20 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Enhancement in axilla | 4 hours after injection
  Hot nodules will be showed in axilla after injection of SENTI-SCINT

CONTACTS AND LOCATIONS:
Overall Officials: Halil KARA, Principal Investigator — Acibadem University
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Sariyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Intra M, Veronesi P, Gentilini OD, Trifiro G, Berrettini A, Cecilio R, Colleoni M, Rietjens M, Luini A, Paganelli G, Veronesi U. Sentinel lymph node biopsy is feasible even after total mastectomy. J Surg Oncol. 2007 Feb 1;95(2):175-9. doi: 10.1002/jso.20670. PMID 17262724
- [Background] Karam A, Stempel M, Cody HS 3rd, Port ER. Reoperative sentinel lymph node biopsy after previous mastectomy. J Am Coll Surg. 2008 Oct;207(4):543-8. doi: 10.1016/j.jamcollsurg.2008.06.139. Epub 2008 Jul 21. PMID 18926457